CLINICAL TRIAL: NCT07384143
Title: Exploring Cognitive Recovery: the Impact of Sensor-based Robotic Rehabilitation in Neurological and Neurodegenerative Disorders
Brief Title: Cognitive Recovery Via Sensor-based Robotic Upper Limb Rehabilitation in Neurological Disorders
Acronym: CROSS-ND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Desiree La Tella, Principal Investigator, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CROSS-ND
Record Dates: First submitted 2025-09-30; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-02

CONDITIONS: PARKINSON DISEASE (Disorder); Multiple Sclerosis; Stroke; Neurological Disorders
MeSH Terms: conditions — Parkinson Disease; Multiple Sclerosis; Stroke; Nervous System Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sensor-Based Robotic Rehabilitation with Cognitive Tasks (SBRR) (Experimental): Participants receive upper limb rehabilitation using sensor-based robotic devices and virtual reality exercises, with integrated cognitive tasks to simultaneously improve motor function and cognitive abilities.
  Interventions: Device: Sensor-Based Robotic Rehabilitation with Cognitive Tasks (SBRR)
- Standard Conventional Therapy (SCT) (Active Comparator): Participants receive conventional upper limb rehabilitation, including standard physiotherapy exercises, without robotic assistance or integrated cognitive tasks.
  Interventions: Device: Standard Conventional Therapy

INTERVENTIONS:
Device: Sensor-Based Robotic Rehabilitation with Cognitive Tasks (SBRR) — Participants receive upper limb rehabilitation using sensor-based robotic devices (e.g., Motore, Armeo Senso, Hand Tutor, Armeo Power, Armeo Spring, Pablo, Amadeo, Diego) combined with virtual reality exercises. The intervention integrates cognitive tasks-such as attention, memory, and executive function exercises-simultaneously with motor training. Therapy is personalized in real-time according to each patient's performance, adjusting difficulty, intensity, and assistance levels to maximize both cognitive and motor recovery.
  Arms: Sensor-Based Robotic Rehabilitation with Cognitive Tasks (SBRR)
Device: Standard Conventional Therapy — Participants receive traditional upper limb rehabilitation, including standard physiotherapy exercises without robotic assistance or integrated cognitive tasks. Therapy focuses on motor recovery using conventional methods, such as repetitive movement exercises, range of motion, and functional tasks, but does not adapt in real-time to patient performance and does not include concurrent cognitive stimulation.
  Arms: Standard Conventional Therapy (SCT)

SUMMARY:
The goal of this clinical trial is to learn if sensor-based robotic upper limb rehabilitation can improve cognitive and motor functions in adults with neurological and neurodegenerative disorders, including Parkinson's disease, multiple sclerosis, and stroke. The main questions it aims to answer are:

Does sensor-based robotic rehabilitation improve cognitive functions such as attention, memory, and executive functions? Does this rehabilitation lead to better motor recovery and daily functioning compared to conventional therapy? Researchers will compare the experimental group receiving robotic rehabilitation with cognitive tasks to the control group receiving conventional therapy to see if the robotic approach leads to greater improvements in both cognitive and motor outcomes.

Participants will:

Receive upper limb rehabilitation using robotic devices and virtual reality-based exercises or conventional therapy Complete a series of neuropsychological assessments before and after the intervention to measure cognitive changes Complete motor function tests before and after the intervention to evaluate physical improvements Participate in 25 training sessions, 2-3 times per week, each lasting 60 minutes

DETAILED DESCRIPTION:
The CROSS-ND study is a randomized controlled trial designed to evaluate the effectiveness of sensor-based robotic upper limb rehabilitation combined with cognitive exercises in adults with neurological and neurodegenerative disorders, including Parkinson's disease, multiple sclerosis, and stroke. Traditional rehabilitation often focuses primarily on motor recovery, but cognitive impairments frequently co-occur and can limit functional gains. This study integrates cognitive tasks within robotic rehabilitation to target both motor and cognitive deficits simultaneously, promoting neuroplasticity and functional independence.

Participants will be randomly assigned to either the experimental group, receiving robotic and virtual reality-based upper limb training with embedded cognitive exercises, or the control group, receiving conventional therapy. Each participant will complete 25 sessions over 2-3 months, with training intensity and difficulty adapted to individual performance.

Assessments will include neuropsychological tests tailored to the patient's condition (ACE-R for Parkinson's, BRB-N for multiple sclerosis, RBANS for stroke) and motor evaluations using standardized tools such as Fugl-Meyer Assessment, Nine Hole Peg Test, and robotic device metrics. Cognitive and motor outcomes will be measured at baseline (T0) and immediately post-intervention (T1).

This study aims to demonstrate that a personalized, integrated rehabilitation approach can improve cognitive functions (attention, memory, executive functions, visuospatial skills) while enhancing motor recovery and daily living activities. Secondary objectives include analyzing correlations between cognitive and motor improvements, evaluating psychological well-being, and exploring the influence of patient characteristics (age, severity, disease stage) on rehabilitation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years;
* FMA-UL 0-31: eligible for exoskeletons and robotic devices with high support. (Armeo Power, Amadeo, Motore)
* FMA-UL 32-47: eligible for end-effectors with medium support. (Armeo Spring, Hand Tutor, Diego)
* FMA-UL 48-52: eligible for sensor-based with low support. (Pablo, Diego, Armeo Senso)
* MoCA: ≤ 20

Exclusion Criteria:

* Severe cognitive disorders
* Behavioral disorders
* Sensory disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2030-02-11 (Estimated); Study Completion 2030-02-11 (Estimated)

PRIMARY OUTCOMES:
Between-group difference in change from baseline in Addenbrooke's Cognitive Examination-Revised (ACE-R) total score (Parkinson's disease) | From baseline (Visit 1) to end of treatment (Visit 2; after completion of 25 rehabilitation sessions; 2-3 sessions/week; each session 60 minutes; total duration ~8-12 weeks).
  Addenbrooke's Cognitive Examination-Revised (ACE-R) total score ranges from 0 to 100, with higher scores indicating better cognitive performance. ACE-R will be administered at baseline (T0) and at end of intervention (T1). The primary metric will be change from baseline (T1 - T0) in ACE-R total score. Results will be summarized as mean (SD) change (or median [IQR] if non-normal) and compared between robotic rehabilitation and conventional therapy groups.
Between-group difference in change from baseline in Brief Repeatable Neuropsychological Test (BRNT) composite score (Multiple Sclerosis) | From baseline (Visit 1) to end of treatment (Visit 2; after completion of 25 rehabilitation sessions; 2-3 sessions/week; each session 60 minutes; total duration ~8-12 weeks).
  The BRB-N is a neuropsychological battery (multiple subtests). Subtest scores will be standardized into z-scores and aggregated into a composite (e.g., mean z-score across predefined subtests). Z-scores have no fixed minimum or maximum; higher values indicate better cognitive performance.The BRNT will be administered at T0 and T1. The primary metric will be change from baseline (T1 - T0) in a composite score derived from BRNT components (standardized z-scores aggregated into a single composite). Results will be summarized as mean (SD) change and compared between groups.
Between-group difference in change from baseline in Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Total Scale Index score (Stroke) | From baseline (Visit 1) to end of treatment (Visit 2; after completion of 25 rehabilitation sessions; 2-3 sessions/week; each session 60 minutes; total duration ~8-12 weeks).
  RBANS Total Scale Index score ranges from 40 to 160, with higher scores indicating better cognitive performance. RBANS will be administered at T0 and T1. The primary metric will be change from baseline (T1 - T0) in RBANS Total Scale Index score. Results will be summarized as mean (SD) change (or median [IQR]) and compared between robotic rehabilitation and conventional therapy groups.

SECONDARY OUTCOMES:
Between-group difference in change from baseline in Fugl-Meyer Assessment-Upper Extremity (FMA-UE/FMA-UL) score | From baseline (T0) to immediately after the final rehabilitation session (T1; after completion of 25 sessions; 2-3 sessions/week; 60 minutes/session; total duration ~8-12 weeks).
  FMA-UE score ranges from 0 to 66, with higher scores indicating better upper-limb motor function. FMA-UL will be assessed at T0 and T1. Metric: change from baseline (T1 - T0). Summaries: mean (SD) change and between-group comparison.
System Usability Scale (SUS) score for robotic device usability at end of treatment | From baseline (T0) to immediately after the final rehabilitation session (T1; after completion of 25 sessions; 2-3 sessions/week; 60 minutes/session; total duration ~8-12 weeks).
  SUS total score ranges from 0 to 100, with higher scores indicating better usability. Participants will complete the SUS at T1 to evaluate usability of the robotic device. Metric: SUS total score. Summaries: mean (SD) (or median [IQR]).
Goal Attainment Scaling (GAS) T-score at end of treatment | From baseline (T0) to immediately after the final rehabilitation session (T1; after completion of 25 sessions; 2-3 sessions/week; 60 minutes/session; total duration ~8-12 weeks).
  GAS is calculated as a standardized T-score typically centered at 50 (SD 10); scores >50 indicate better-than-expected goal attainment, while scores <50 indicate less-than-expected attainment. Individualized rehabilitation goals will be defined at baseline and evaluated at T1 using GAS. Metric: GAS T-score at T1 (or change, se lo calcoli). Summaries: mean (SD) and between-group comparison.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Centro Neurolesi Bonino-Pulejo, Messina, Maine, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bard-Pondarré R, Villepinte C, Roumenoff F, Lebrault H, Bonnyaud C, Pradeau C, Bensmail D, Isner-Horobeti ME, Krasny-Pacini A. Goal Attainment Scaling in rehabilitation: An educational review providing a comprehensive didactical tool box for implementing Goal Attainment Scaling. J Rehabil Med. 2023 Jun 14;55:jrm6498. doi: 10.2340/jrm.v55.6498. PMID: 37317629; PMCID: PMC10301855.
- [Background] Moulaei K, Moulaei R, Bahaadinbeigy K. The most used questionnaires for evaluating the usability of robots and smart wearables: A scoping review. Digit Health. 2024 Apr 9;10:20552076241237384. doi: 10.1177/20552076241237384. PMID: 38601185; PMCID: PMC11005511.
- [Background] Bull R, Espy KA, Senn TE. A comparison of performance on the Towers of London and Hanoi in young children. J Child Psychol Psychiatry. 2004 May;45(4):743-54. doi: 10.1111/j.1469-7610.2004.00268.x. PMID: 15056306.
- [Background] Randolph C, Tierney MC, Mohr E, Chase TN. The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS): preliminary clinical validity. J Clin Exp Neuropsychol. 1998 Jun;20(3):310-9. doi: 10.1076/jcen.20.3.310.823. PMID 9845158
- [Background] Solari A, Filippini G, Mendozzi L, Ghezzi A, Cifani S, Barbieri E, Baldini S, Salmaggi A, Mantia LL, Farinotti M, Caputo D, Mosconi P. Validation of Italian multiple sclerosis quality of life 54 questionnaire. J Neurol Neurosurg Psychiatry. 1999 Aug;67(2):158-62. doi: 10.1136/jnnp.67.2.158. PMID 10406981
- [Background] Tedone N, Vizzino C, Meani A, Gallo A, Altieri M, D'Ambrosio A, Pantano P, Piervincenzi C, Tommasin S, De Stefano N, Cortese R, Stromillo ML, Rocca MA; INNI network; Filippi M. The brief repeatable battery of neuropsychological tests (BRB-N) version a: update of Italian normative data from the Italian Neuroimaging Network Initiative (INNI). J Neurol. 2024 Apr;271(4):1813-1823. doi: 10.1007/s00415-023-12108-z. Epub 2023 Dec 7. PMID: 38060030.
- [Background] Galeoto G, Colalelli F, Massai P, Berardi A, Tofani M, Pierantozzi M, Servadio A, Fabbrini A, Fabbrini G. Quality of life in Parkinson's disease: Italian validation of the Parkinson's Disease Questionnaire (PDQ-39-IT). Neurol Sci. 2018 Nov;39(11):1903-1909. doi: 10.1007/s10072-018-3524-x. Epub 2018 Aug 7. PMID 30088166
- [Background] Nocentini, U., Giordano, A., Vincenzo, S. D., Panella, M., & Pasqualetti, P. (2006). The Symbol Digit Modalities Test--Oral version: Italian normative data. Functional neurology, 21(2), 93-96.
- [Background] Siciliano M, Chiorri C, Battini V, Sant'Elia V, Altieri M, Trojano L, Santangelo G. Regression-based normative data and equivalent scores for Trail Making Test (TMT): an updated Italian normative study. Neurol Sci. 2019 Mar;40(3):469-477. doi: 10.1007/s10072-018-3673-y. Epub 2018 Dec 7. PMID 30535956
- [Background] Siciliano M, Raimo S, Tufano D, Basile G, Grossi D, Santangelo F, Trojano L, Santangelo G. The Addenbrooke's Cognitive Examination Revised (ACE-R) and its sub-scores: normative values in an Italian population sample. Neurol Sci. 2016 Mar;37(3):385-92. doi: 10.1007/s10072-015-2410-z. Epub 2015 Nov 12. PMID 26563847
- [Background] Hoonhorst MH, Nijland RH, van den Berg JS, Emmelot CH, Kollen BJ, Kwakkel G. How Do Fugl-Meyer Arm Motor Scores Relate to Dexterity According to the Action Research Arm Test at 6 Months Poststroke? Arch Phys Med Rehabil. 2015 Oct;96(10):1845-9. doi: 10.1016/j.apmr.2015.06.009. Epub 2015 Jul 2. PMID: 26143054.
- [Background] Li, X., Tang, Z., Wu, D., Su, L., Zheng, Y., Chen, P., Zhang, Y., Dou, Z., Li, K., & Hoseinbeyki, A. (2021). Analysis of the Positive Effect of Robot-Assisted Virtual Reality Technology on Rehabilitation of Motor Function and Nerve Function in Cerebral Stroke Patients. J. Medical Imaging Health Informatics, 11, 595-600. https://doi.org/10.1166/jmihi.2021.3372.
- [Background] Manuli A, Maggio MG, Latella D, Cannavo A, Balletta T, De Luca R, Naro A, Calabro RS. Can robotic gait rehabilitation plus Virtual Reality affect cognitive and behavioural outcomes in patients with chronic stroke? A randomized controlled trial involving three different protocols. J Stroke Cerebrovasc Dis. 2020 Aug;29(8):104994. doi: 10.1016/j.jstrokecerebrovasdis.2020.104994. Epub 2020 Jun 13. PMID 32689601
- [Background] Metzger JC, Lambercy O, Califfi A, Conti FM, Gassert R. Neurocognitive robot-assisted therapy of hand function. IEEE Trans Haptics. 2014 Apr-Jun;7(2):140-9. doi: 10.1109/TOH.2013.72. PMID 24968378
- [Background] Calabrò RS, Naro A, Russo M, Bramanti P, Carioti L, Balletta T, et al.. Shaping neuroplasticity by using powered exoskeletons in patients with stroke: a randomized clinical trial. J Neuroeng Rehabil. (2018) 15:35. 10.1186/s12984-018-0377-8
- [Background] Kiper P, Richard M, Stefanutti F, Pierson-Poinsignon R, Cacciante L, Perin C, Mazzucchelli M, Vigano B, Meroni R. Combined Motor and Cognitive Rehabilitation: The Impact on Motor Performance in Patients with Mild Cognitive Impairment. Systematic Review and Meta-Analysis. J Pers Med. 2022 Feb 14;12(2):276. doi: 10.3390/jpm12020276. PMID 35207764
- [Background] Riener R, Lunenburger L, Colombo G. Human-centered robotics applied to gait training and assessment. J Rehabil Res Dev. 2006 Aug-Sep;43(5):679-94. doi: 10.1682/jrrd.2005.02.0046. PMID 17123208
- [Background] Aprile I, Guardati G, Cipollini V, Papadopoulou D, Monteleone S, Redolfi A, Garattini R, Sacella G, Noro F, Galeri S, Carrozza MC, Germanotta M. Influence of Cognitive Impairment on the Recovery of Subjects with Subacute Stroke Undergoing Upper Limb Robotic Rehabilitation. Brain Sci. 2021 Apr 30;11(5):587. doi: 10.3390/brainsci11050587. PMID 33946452
- [Background] Aprile I, Guardati G, Cipollini V, Papadopoulou D, Mastrorosa A, Castelli L, Monteleone S, Redolfi A, Galeri S, Germanotta M. Robotic Rehabilitation: An Opportunity to Improve Cognitive Functions in Subjects With Stroke. An Explorative Study. Front Neurol. 2020 Nov 19;11:588285. doi: 10.3389/fneur.2020.588285. eCollection 2020. PMID 33329334
- [Background] Mehrholz, J., Pollock, A., Pohl, M. et al. Systematic review with network meta-analysis of randomized controlled trials of robotic-assisted arm training for improving activities of daily living and upper limb function after stroke. J NeuroEngineering Rehabil 17, 83 (2020). https://doi.org/10.1186/s12984-020-00715-0
- [Background] Xie H, Li X, Huang W, Yin J, Luo C, Li Z, Dou Z. Effects of robot-assisted task-oriented upper limb motor training on neuroplasticity in stroke patients with different degrees of motor dysfunction: A neuroimaging motor evaluation index. Front Neurosci. 2022 Sep 16;16:957972. doi: 10.3389/fnins.2022.957972. PMID: 36188465; PMCID: PMC9523102.
- [Background] Calabrò RS, Morone G, Naro A, Gandolfi M, Liotti V, D'aurizio C, Straudi S, Focacci A, Pournajaf S, Aprile I, Filoni S, Zanetti C, Leo MR, Tedesco L, Spina V, Chisari C, Taveggia G, Mazzoleni S, Smania N, Paolucci S, Franceschini M, Bonaiuti D. Robot-Assisted Training for Upper Limb in Stroke (ROBOTAS): An Observational, Multicenter Study to Identify Determinants of Efficacy. J Clin Med. 2021 Nov 11;10(22):5245. doi: 10.3390/jcm10225245. PMID: 34830527; PMCID: PMC8622640
- [Background] Germanotta M, Cortellini L, Insalaco S, Aprile I. Effects of Upper Limb Robot-Assisted Rehabilitation Compared with Conventional Therapy in Patients with Stroke: Preliminary Results on a Daily Task Assessed Using Motion Analysis. Sensors (Basel). 2023 Mar 13;23(6):3089. doi: 10.3390/s23063089. PMID 36991799
- [Background] Zengin-Metli D, Ozbudak-Demir S, Eraktas I, Binay-Safer V, Ekiz T. Effects of robot assistive upper extremity rehabilitation on motor and cognitive recovery, the quality of life, and activities of daily living in stroke patients. J Back Musculoskelet Rehabil. 2018;31(6):1059-1064. doi: 10.3233/BMR-171015. PMID 29966188
- [Background] Adomavičiene A, Daunoravičiene K, Kubilius R, VarŽaityte L, Raistenskis J. Influence of new technologies on post-stroke rehabilitation: a comparison of Armeo spring to the kinect system. Med. (2019) 55:98. 10.3390/medicina55040098.
- [Background] Bui KD, Johnson MJ. Robot-based measures of upper limb cognitive-motor interference across the HIV-stroke spectrum. In: IEEE International Conference on Rehabilitation Robotics. (2019) p. 530-5.
- [Background] Chen C, Leys D, Esquenazi A. The interaction between neuropsychological and motor deficits in patients after stroke. Neurology. 2013 Jan 15;80(3 Suppl 2):S27-34. doi: 10.1212/WNL.0b013e3182762569. PMID 23319483
- [Background] Lamb F, Anderson J, Saling M, Dewey H. Predictors of subjective cognitive complaint in postacute older adult stroke patients. Arch Phys Med Rehabil. 2013 Sep;94(9):1747-52. doi: 10.1016/j.apmr.2013.02.026. Epub 2013 Mar 22. PMID 23529143
- [Background] Pollock A, Farmer SE, Brady MC, Langhorne P, Mead GE, Mehrholz J, van Wijck F. Interventions for improving upper limb function after stroke. Cochrane Database Syst Rev. 2014 Nov 12;2014(11):CD010820. doi: 10.1002/14651858.CD010820.pub2. PMID 25387001
- [Background] Pendlebury ST, Rothwell PM. Prevalence, incidence, and factors associated with pre-stroke and post-stroke dementia: a systematic review and meta-analysis. Lancet Neurol. 2009 Nov;8(11):1006-18. doi: 10.1016/S1474-4422(09)70236-4. Epub 2009 Sep 24. PMID 19782001
- [Background] Gottesman RF, Hillis AE. Predictors and assessment of cognitive dysfunction resulting from ischaemic stroke. Lancet Neurol. 2010 Sep;9(9):895-905. doi: 10.1016/S1474-4422(10)70164-2. PMID 20723846
- [Background] Lesniak M, Bak T, Czepiel W, Seniow J, Czlonkowska A. Frequency and prognostic value of cognitive disorders in stroke patients. Dement Geriatr Cogn Disord. 2008;26(4):356-63. doi: 10.1159/000162262. Epub 2008 Oct 14. PMID 18852488
- [Background] Nys GM, van Zandvoort MJ, de Kort PL, van der Worp HB, Jansen BP, Algra A, de Haan EH, Kappelle LJ. The prognostic value of domain-specific cognitive abilities in acute first-ever stroke. Neurology. 2005 Mar 8;64(5):821-7. doi: 10.1212/01.WNL.0000152984.28420.5A. PMID 15753416
- [Background] Loetscher T, Potter KJ, Wong D, das Nair R. Cognitive rehabilitation for attention deficits following stroke. Cochrane Database Syst Rev. 2019 Nov 10;2019(11):CD002842. doi: 10.1002/14651858.CD002842.pub3. PMID 31706263

DOCUMENTS (2):
  • Study Protocol (2025-01-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT07384143/Prot_000.pdf
  • Informed Consent Form (2025-01-24): https://cdn.clinicaltrials.gov/large-docs/43/NCT07384143/ICF_001.pdf